CLINICAL TRIAL: NCT01694225
Title: Estimating the Adherence Rate of a Monthly Bubble Package Among Patients Prescribed Adjuvant Endocrine Therapy in Breast Cancer Survivors
Brief Title: Adherence Rate of Monthly Bubble Package Among Patients Prescribed Adjuvant Endocrine Therapy in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Elizabeth Riley, Associate Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BCC-BRE-12-Adherence
Record Dates: First submitted 2012-09-23; First posted 2012-09-27 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Anti-estrogen therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bubble package for monthly prescription (Experimental): use of bubble packaging for monthly prescription
  Interventions: Other: bubble packaging for monthly prescription

INTERVENTIONS:
Other: bubble packaging for monthly prescription — Monthly bubble packaging among women prescribed anti-estrogens

SUMMARY:
This study aims to establish the feasibility of using a monthly bubble package to improve compliance rates among women prescribed adjuvant endocrine therapy.

DETAILED DESCRIPTION:
This study uses Bubble packaging to provide a cost effective way to improve compliance and help direct further interventions to ensure adherence in women on anti-estrogen therapy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Estrogen receptor positive (> 1% estrogen expression) by immunohistochemistry
* Invasive breast cancer (stage I, II, III) or DCIS considered for adjuvant endocrine therapy

Exclusion Criteria:

* Patients with metastatic disease (stage IV)
* Patients less than 18 years of age
* Prisoners
* Patients are unable to fill prescriptions at the BCC pharmacy due to insurance limitations or personal preference

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-07; Primary Completion 2018-01-28 (Actual); Study Completion 2018-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Riley, MD, Principal Investigator — James Graham Brown Cancer Center- U of Louisville
Locations (1):
- James Graham Brown Cancer Center-University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
no plan for public sharing of individual participant data